CLINICAL TRIAL: NCT02281578
Title: Community-based Combination HIV Prevention in Tanzanian Women at Heightened Risk
Brief Title: Community-based Combination HIV Prevention in Tanzanian Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Principal Investigator, Deanna Kerrigan, Associate Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: R01MH104044 (NIH)
Record Dates: First submitted 2014-10-29; First posted 2014-11-03 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: HIV
Keywords: Sex Workers; Prevention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination prevention (Experimental): Community-based, combination HIV prevention intervention package
  Interventions: Behavioral: Community-based combination HIV prevention intervention
- Standard of care (Active Comparator): Locally run standard of care HIV prevention, treatment and care services
  Interventions: Behavioral: Standard of care HIV services

INTERVENTIONS:
Behavioral: Community-based combination HIV prevention intervention — The combination package will include integrated biomedical, behavioral and structural components: (1) mobile HIV testing and risk reduction counseling; (2) service navigation to facilitate access to treatment and retention in care; (3) sensitivity training for HIV clinical care providers; (4) SMS text messages to promote adherence to care and ART; (5) venue-based peer education and condom distribution; and (6) a community drop-in-center to promote cohesion and collective action to reduce stigma and discrimination.
  Arms: Combination prevention
Behavioral: Standard of care HIV services — Locally available standard of care HIV prevention, treatment and care services
  Arms: Standard of care

SUMMARY:
The Phase II trial will assess the feasibility, acceptance, safety, pathways, and initial effectiveness of a community-based combination HIV prevention intervention among bar-based female sex workers in Iringa, Tanzania. Results will inform an appropriately powered Phase III RCT as warranted.

DETAILED DESCRIPTION:
Combination HIV prevention demonstrates significant promise in reducing burden of disease. To maximize its effectiveness combination prevention must be tailored to a given context and population. From the beginning of the global HIV epidemic, female sex workers (FSWs) have been found to be at heightened risk for infection. More recently the role that sex work plays in ongoing HIV transmission dynamics has been more clearly established in generalized epidemics, where previously limited attention was paid to the role of key populations. The greater vulnerability of FSWs is now widely understood to be associated with social and structural factors including the intense stigma, discrimination and violence they often face and the unsafe environments in which they live and work. These factors are known to limit both protective sexual behaviors and engagement in HIV testing, care and treatment services. Comprehensive, community-based HIV prevention approaches addressing the aforementioned social and structural vulnerabilities to HIV infection among FSWs have been shown to be effective in South Asia and in Latin America. However, in sub-Saharan Africa where the impact of HIV is the greatest, no systematic efforts to develop and evaluate the feasibility and effectiveness of community-based combination HIV prevention among FSWs has occurred.

The investigators will conduct a two-arm Phase II community randomized controlled trial of a community-based combination HIV prevention intervention among FSWs in Iringa, Tanzania. The model was developed on the basis of prior formative research and mapping and utilizes an ongoing research infrastructure. The combination package will include integrated biomedical, behavioral and structural components: (1) mobile HIV testing and risk reduction counseling; (2) service navigation to facilitate access to treatment and retention in care; (3) sensitivity training for HIV clinical care providers; (4) SMS text messages to promote adherence to care and ART; (5) venue-based peer education and condom distribution; and (6) a community drop-in-center to promote cohesion and collective action to reduce stigma and discrimination. The investigators seek to establish base rates of key outcomes including HIV incidence and viral load suppression, examine the socio-structural and behavioral pathways of the intervention, assess feasibility, acceptability and safety, and document preliminary effectiveness. Should compelling indications of safety, feasibility, acceptability and initial effectiveness be found, study results will inform the first Phase III RCT of community-based combination HIV prevention among FSWs.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old, female, exchange sex for money in entertainment venue
2. key informants working on HIV among sex workers in the region.

Exclusion Criteria:

* Psychiatric/psychological condition impeding informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
HIV incidence | 18 months
  Biologic assessment of new infections among HIV-uninfected participants via blood draw
Viral load suppression | 18 months
  Biological assessment of viral suppression among HIV-infected participants via blood draw

SECONDARY OUTCOMES:
Consistent condom use | 18 months
  Consistent condom use with clients among all participants via survey measures
Adherence to ART | 18 months
  Adherence to ART medication among those living with HIV via survey measures

CONTACTS AND LOCATIONS:
Overall Officials: Deanna L Kerrigan, PhD, MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- MUHAS, Iringa, Tanzania

REFERENCES:
- [Background] Kerrigan D, Mbwambo J, Likindikoki S, Davis W, Mantsios A, Beckham SW, Leddy A, Shembilu C, Mwampashi A, Aboud S, Galai N. Project Shikamana: Community Empowerment-Based Combination HIV Prevention Significantly Impacts HIV Incidence and Care Continuum Outcomes Among Female Sex Workers in Iringa, Tanzania. J Acquir Immune Defic Syndr. 2019 Oct 1;82(2):141-148. doi: 10.1097/QAI.0000000000002123. PMID 31513552
- [Background] Kerrigan D, Mbwambo J, Likindikoki S, Beckham S, Mwampashi A, Shembilu C, Mantsios A, Leddy A, Davis W, Galai N. Project Shikamana: Baseline Findings From a Community Empowerment-Based Combination HIV Prevention Trial Among Female Sex Workers in Iringa, Tanzania. J Acquir Immune Defic Syndr. 2017 Jan 1;74 Suppl 1(Suppl 1):S60-S68. doi: 10.1097/QAI.0000000000001203. PMID 27930613
- [Derived] Beckham SW, Mantsios A, Galai N, Likindikoki S, Mbwambo J, Davis W, Kerrigan D. Acceptability of multiple modalities of pre-exposure prophylaxis (PrEP) among female sex workers in Tanzania: a mixed-methods study. BMJ Open. 2022 Aug 17;12(8):e058611. doi: 10.1136/bmjopen-2021-058611. PMID 35977762